CLINICAL TRIAL: NCT00825799
Title: Validation of Serum Markers as a Bioassay for Unipolar Depression
Brief Title: Serum Markers as a Bioassay for Unipolar Depression
Status: Completed | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: Ridge Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 00435
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-06

CONDITIONS: Major Depression
Keywords: biomarker; depression; blood test
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Major Depressive Disorder: Adults with major depressive disorder who are experiencing a current depressive episode.
- Healthy controls: Individuals without any Axis I psychiatric diagnosis who are matched to depressed subjects by age and sex.

SUMMARY:
The goal of the study is to validate a biomarker assay for unipolar depression based on serum proteins involved in inflammation, metabolism, and stress response. The study will compare patients with a current major depressive episode to individuals with no history of depression. The hypothesis is that the assay can serve as a diagnostic tool that would be more objective than standard diagnostic questionnaires.

ELIGIBILITY:
Inclusion Criteria (Depressed):

* Aged 18 to 60.
* Meets DSM-IV criteria for Unipolar Major Depression, either single or recurrent.
* 21 item Hamilton Depression rating scale score greater than 18.
* Capable of providing informed consent.
* Has an established residence and phone number.

Exclusion Criteria:

* Meets DSM-IV criteria for Bipolar Disorder, Schizophrenia, Schizoaffective disorder or other major Axis I Psychiatric disorders (except for depression and phobia per above).
* Addison's Disease, Cushing's Disease, or other known dysfunction of the HPA-cortisol axis.
* Rheumatoid arthritis, lupus, or other condition associated with increased inflammation.
* Regular use of non-steroidal anti-inflammatory medications, steroids, or other medications know to interact with the inflammatory process of the HPA axis.
* A medical condition or regular use of a mediation, which I the opinion of the investigator is likely to influence the inflammatory or HPA responses.
* Pregnancy.
* Meets DSM-IV criteria for substance abuse or dependence in the last month.
* Regular cigarette smoking.
* History of fainting or other significant adverse event during blood drawing in the past.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are recruited from the community by advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Protein biomarker MDDScore. | 0 weeks

SECONDARY OUTCOMES:
Score on Hamilton Depression Rating Scale (HDRS). | 0 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Henry, MD, Principal Investigator — Steward St. Elizabeth's Medical Center
Locations (1):
- Steward St. Elizabeth's Medical Center, Boston, Massachusetts, United States